CLINICAL TRIAL: NCT07078019
Title: Estimation of Pain Level in Patients With Chronic Low Back Pain From Voice Recordings: A Comparative Pilot Study With VAS and Lumbar Function Index
Brief Title: Predicting Pain and Disability From Voice Recordings in Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: nurmuhammet tas (Other Government)
Collaborators: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, nurmuhammet tas, Principal Investigator, Erzurum Regional Training & Research Hospital
Organization: Erzurum Regional Training & Research Hospital (Other Government)
Other Study IDs: erzurum rtrh4
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Chronic low back pain; Voice analysis; Oswestry Disability Index; Roland-Morris Questionnaire; Acoustic biomarkers; Pain assessment; VAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- VAS 0 Group: Participants with chronic low back pain reporting a VAS score of 0
  Interventions: Other: Voice Recording Procedure
- VAS 1 Group: Participants with chronic low back pain reporting a VAS score of 1
  Interventions: Other: Voice Recording Procedure
- VAS 2 Group: Participants with chronic low back pain reporting a VAS score of 2
  Interventions: Other: Voice Recording Procedure
- VAS 3 Group: Participants with chronic low back pain reporting a VAS score of 3
  Interventions: Other: Voice Recording Procedure
- VAS 4 Group: Participants with chronic low back pain reporting a VAS score of 4
  Interventions: Other: Voice Recording Procedure
- VAS 5 Group: Participants with chronic low back pain reporting a VAS score of 5
  Interventions: Other: Voice Recording Procedure
- VAS 6 Group: Participants with chronic low back pain reporting a VAS score of 6
  Interventions: Other: Voice Recording Procedure
- VAS 7 Group: Participants with chronic low back pain reporting a VAS score of 7
  Interventions: Other: Voice Recording Procedure
- VAS 8 Group: Participants with chronic low back pain reporting a VAS score of 8
  Interventions: Other: Voice Recording Procedure
- VAS 9 Group: Participants with chronic low back pain reporting a VAS score of 9
  Interventions: Other: Voice Recording Procedure
- VAS 10 Group: Participants with chronic low back pain reporting a VAS score of 10
  Interventions: Other: Voice Recording Procedure

INTERVENTIONS:
Other: Voice Recording Procedure — Participants will be asked to read a standardized one-minute text aloud in a quiet room. Their voices will be recorded using a high-quality microphone. The recordings will later be analyzed for acoustic features such as pitch, speech rate, pauses, and intonation.
  This procedure is non-invasive and does not involve any clinical or pharmacological intervention.

SUMMARY:
This study aims to investigate whether pain intensity (assessed by Visual Analog Scale - VAS) and functional impairment (Roland-Morris Disability Questionnaire [RMDQ] or Oswestry Disability Index [ODI]) in patients with chronic low back pain can be estimated using acoustic features extracted from short voice recordings.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most common musculoskeletal complaints and a leading cause of disability worldwide. Assessing pain severity and its impact on function is primarily reliant on self-reported tools such as the Visual Analog Scale (VAS) and functional indices like the Oswestry Disability Index (ODI) or Roland-Morris Disability Questionnaire (RMDQ). However, these tools may be influenced by subjectivity and reporting bias. Therefore, objective and non-invasive methods for pain assessment are needed.

This pilot observational study aims to investigate whether acoustic characteristics of voice recordings can be used to estimate pain intensity and functional impairment in individuals with CLBP. The hypothesis is that pain-induced changes in a patient's psychophysiological state may alter specific voice parameters (e.g., pitch, speech rate, pauses, intonation), which can be quantified through acoustic analysis.

After obtaining ethical approval, data will be collected at the Department of Physical Medicine and Rehabilitation. A total of 110 participants aged 18-70 years with chronic low back pain will be recruited. Each participant will be asked to read a standardized one-minute text aloud, and their voice will be recorded in a controlled setting. On the same day, participants will complete the VAS and either the ODI or RMDQ questionnaires.

Voice recordings will be analyzed using speech signal processing tools to extract features such as fundamental frequency, speech rate, articulation rate, pauses, and prosodic variations. These voice parameters will then be statistically correlated with VAS and disability scores.

Participants will be grouped by their VAS score (0-10), with an equal number of participants targeted for each pain level to ensure balanced data distribution. Written and verbal informed consent will be obtained from all participants. All recordings and data will be anonymized, and participants will retain the right to withdraw from the study at any time without consequence.

This study adheres to the principles of the Declaration of Helsinki and aims to provide early evidence supporting the feasibility of voice-based pain assessment. If successful, this approach could pave the way for low-cost, scalable, and objective tools to assist in the diagnosis and monitoring of chronic pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Diagnosed with chronic low back pain and attending the physical medicine and rehabilitation clinic
* Literate (able to read and write)

Exclusion Criteria:

* Age below 18
* Illiterate individuals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 70 years with chronic low back pain who are literate and visiting the physical medicine and rehabilitation outpatient clinic. Participants must be able to read and speak Turkish fluently to complete questionnaires and perform the standardized reading task for voice recording. Individuals with acute back pain, neurological disorders, or communication impairments are excluded.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between voice features and pain level (VAS score) | At the time of enrollment
  Voice parameters such as pitch, tone, speech rate, and pauses will be analyzed and statistically correlated with pain levels as measured by the Visual Analog Scale (VAS).
  The VAS is a self-reported pain measurement tool scored on a scale from 0 to 10, where:
  0 indicates no pain, and
  10 indicates the worst pain imaginable. Higher scores represent worse pain outcomes.

SECONDARY OUTCOMES:
Correlation between voice features and functional impairment (Oswestry Disability Index [ODI] or Roland-Morris Disability Questionnaire [RMDQ]) | At the time of enrollment
  Functional disability levels will be assessed using either the Oswestry Disability Index (ODI) or the Roland-Morris Disability Questionnaire (RMDQ) and will be correlated with acoustic voice features such as pitch, tone, speech rate, and pauses.
  The ODI is scored from 0 to 100, with higher scores indicating greater disability.
  The RMDQ is scored from 0 to 24, where higher scores also indicate greater disability.

IPD SHARING:
Plan to Share IPD: No
Anonymized data may be used in aggregated form for publication.